CLINICAL TRIAL: NCT03108820
Title: Collaborative Care for the Older Injured Patient: A Trauma Medical Home
Brief Title: Trauma Medical Home for Older Injured Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Northwestern University (Other); University of Missouri, Kansas City (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Ben Zarzaur, MD, MPH, Associate Professor of Surgery, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1612690852; 1R01AG052493-01A1 (NIH)
Record Dates: First submitted 2017-04-06; First posted 2017-04-11 (Actual); Results first posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TMH Intervention (Experimental): The multidisciplinary team which develops and carries out the intervention includes a care coordinator who will organize and align recovery resources, a Trauma Surgeon (Dr. Zarzaur), a critical care physician (Dr. Khan), a geriatrician with expertise in collaborative care (Dr. Boustani), and an ICU collaborative care nurse (Dr. Lasiter). Using the Healthy Aging Brain Care monitor, care protocols, specialized software, and specific care protocols, the multidisciplinary team will modulate the intensity and the type of intervention the patient's receive based on the patient's needs. The intervention will last from the time of discharge to 6 months after injury.
  Interventions: Behavioral: TMH Intervention
- Usual Care (Active Comparator): Review hospital discharge and rehabilitation plan, identify the primary care physician responsible for the patient care. Patients will receive education on communication skills; caregiver coping skills; and legal and financial advice. Patients randomized to usual care will receive no further interventions.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: TMH Intervention — Home visits and close interaction with injured patient to assure plan for care is being followed.
  Arms: TMH Intervention
Other: Usual Care — Review hospital discharge and rehabilitation plan, identification of primary care provider, provision of educational materials on communication skills, caregiver coping skills, and legal and financial advice.
  Arms: Usual Care

SUMMARY:
This proposal aims to conduct a randomized controlled trial to evaluate the efficacy of a 6-month collaborative care intervention in improving the functional and psychological recovery of 430 injury survivors 50 and older. The trial has the following specific aims: 1) Evaluate the ability of the TMH intervention to improve the physical recovery of older injury survivors; and 2) Evaluate the ability of the TMH intervention to improve the psychological recovery of older injury survivors; and 3) Evaluate the ability of the TMH intervention to reduce healthcare costs of older injury survivors and evaluate the cost of effectiveness of the TMH intervention.

DETAILED DESCRIPTION:
Despite the potential for full recovery surprisingly few older injury survivors are able to realize maximal recovery of function and quality of life after injury due to fragmentation of care delivery and lack of focus on psychological symptoms in the early post-injury period. Older injured adults are at particular risk of death and disability after injury. Thus, a fundamental gap in knowledge exists regarding the best way to enhance the recovery of injury survivors. The continued existence of this gap is an important problem because unless it is filled, injury survivors will continue to suffer from potentially reversible impairments of health and well-being. The long-term goal of this line of research is to improve the health and quality of care for injured patients. Indiana University School of Medicine researchers have over 20 years of experience developing innovative and effective collaborative care models that integrate with primary care and specialty physicians to address the complex biopsychosocial needs of patients with chronic disease states, such as dementia and depression. Based on these successes, an interdisciplinary team of clinical investigators at Indiana University revised the collaborative care model to meet the needs of injury survivors who are in an active recovery state. This injury specific collaborative care model is called the Trauma Medical Home (TMH). This proposal aims to conduct a randomized controlled trial to evaluate the efficacy of a 6-month collaborative care intervention in improving the functional and psychological recovery of 430 injury survivors 50 and older. The trial has the following specific aims: 1) Evaluate the ability of the TMH intervention to improve the physical recovery of older injury survivors; and 2) Evaluate the ability of the TMH intervention to improve the psychological recovery of older injury survivors; and 3) Evaluate the ability of the TMH intervention to reduce healthcare costs of older injury survivors and evaluate the cost of effectiveness of the TMH intervention. The research proposed in this application is innovative, in our opinion, because it represents a new and substantive departure from the status quo. Previous collaborative care models focused on chronic care management and they lack rapid adaptability. Because the recovery trajectory of injured patients is dynamic and changes quickly, the innovations in this proposal have to do with providing real-time feedback to a care coordinator that will allow the care coordinator to adjust an injury specific collaborative care protocol to meet the needs of the injured as they move through the dynamic recovery period after injury. This contribution will be significant as broad application of the Trauma Medical Home in trauma centers and trauma systems nationwide could result in better health and improved quality of post-injury care for older injured patients. Improved physical health and fewer psychological symptoms, will likely result in better overall functional ability, the increased ability to return to work and less reliance on family, social, and health care resources.

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking adult age 50 years and older;
2. admitted to Indiana University Health - Methodist or Eskenazi Health hospitals;
3. able to provide consent or has a legally authorized representative to provide consent;
4. access to a telephone;
5. and an injury severity score (ISS) of 9 or greater.

Exclusion Criteria:

1. have a self-reported diagnosis of cancer with short life expectancy;
2. have a history of dementing illnesses and other neurodegenerative disease such as Alzheimer disease, Parkinson disease, or vascular dementia;
3. have a significant traumatic brain injury (defined as the presence of any intracranial blood on Computed Tomography scan of the head or best Glasgow Coma Scale Score of less than 13 at the time of study enrollment);
4. have any spinal cord injury with persistent neurologic deficit at the time of study enrollment;
5. are pregnant women (assessed by a urine pregnancy test);
6. have a primary residence outside the state of Indiana;
7. are incarcerated at the time of study enrollment;
8. have an acute stroke upon admission or develop a stroke as a new event during the course of hospitalization;
9. unable to complete study questionnaire due to severe hearing loss;
10. recent history of alcohol or substance abuse;
11. discharged to a permanent care facility;
12. admitted with a burn affecting >10% total body surface area.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ben Zarzaur, MD, MPH, Principal Investigator — University of Wisconsin, Madison
Locations (4):
- United States (4):
  - Eskenazi Hospital, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - St. Vincent Indianapolis, Indianapolis, Indiana
  - UW Health - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zarzaur BL, Holler E, Ortiz D, Perkins A, Lasiter S, Gao S, French DD, Khan B, Boustani M. Collaborative Care for Injured Older Adults: The Trauma Medical Home Randomized Clinical Trial. JAMA Surg. 2024 Jul 1;159(7):756-764. doi: 10.1001/jamasurg.2024.1043. PMID 38717762
- [Derived] Ortiz D, Meagher AD, Lindroth H, Holler E, Gao S, Khan B, Lasiter S, Boustani M, Zarzaur B. A trauma medical home, evaluating collaborative care for the older injured patient: study protocol for a randomized controlled trial. Trials. 2020 Jul 16;21(1):655. doi: 10.1186/s13063-020-04582-x. PMID 32678026

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TMH Intervention | Usual Care
Started | 216 | 214 (1 withdrew immediately after randomization so 213 and was not included in the analysis.)
6 Month Assessment | 158 | 166
Completed | 148 | 151
Not Completed | 68 | 63
Not completed — Lost to Follow-up | 30 | 28
Not completed — Withdrawal by Subject | 32 | 24
Not completed — Death | 6 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TMH Intervention | Usual Care | Total
Number analyzed (Participants) | 216 | 213 | 429
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (10.9) | 68.9 (10.6) | 69.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 114 | 228
  Male | 102 | 99 | 201
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 19 | 18 | 37
  Race: Other | 2 | 2 | 4
  Race: White | 195 | 193 | 388
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic | 2 | 1 | 3
  Ethnicity: Non-Hispanic | 214 | 212 | 426
Region of Enrollment [Number; unit: participants]
  United States | 216 | 213 | 429
Mechanism of Injury [Count of Participants; unit: Participants]
  Fall | 121 | 122 | 243
  Motor Vehicle Crash | 66 | 66 | 132
  Other | 29 | 25 | 54
Injury Severity Score [Mean (Standard Deviation); unit: score] — The Injury Severity Score (ISS) is measured on a scale of 1-75 with higher scores associated with an increased probability of mortality. Scores of more than 9 are considered moderate to severe injury.
  score | 12 (3.9) | 12.5 (5.1) | 12.3 (4.6)
Hospital Length of Stay [Median (Inter-Quartile Range); unit: days] | 7 [4 to 10] | 6 [4 to 10] | 7 [4 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Change in Self Reported Physical Recovery
Description: As determined using the Physical Component Score of Short form (SF) SF-36. Score range: 0-100, higher scores indicate a better health state. The change is between baseline and 12 months.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMH Intervention | Usual Care
Number analyzed (Participants) | 148 | 151
score on a scale | 40.42 (12.82) | 39.18 (12.43)

2. Primary Outcome: Change in Physical Recovery
Description: As determined using the Short Physical Performance Battery (SPPB). SPPB total score ranges from 0 (worst performance) to 12 points (best performance). The change was determined between baseline and 12 months.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMH Intervention | Usual Care
Number analyzed (Participants) | 71 | 65
score on a scale | 8.28 (3.88) | 8.00 (3.60)

3. Primary Outcome: Change in Self Reported Psychological Recovery
Description: As determined using the Mental Component Score of SF-36. Score range: 0-100, higher scores indicate a better health state. The change was determined between baseline and 12 months.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMH Intervention | Usual Care
Number analyzed (Participants) | 148 | 151
score on a scale | 53.92 (10.02) | 53.21 (10.82)

4. Primary Outcome: Healthcare Utilization
Description: As determined by hospital readmission
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | TMH Intervention | Usual Care
Number analyzed (Participants) | 216 | 213
Participants
  Readmission within 1 year | 70 | 71
  No readmission | 146 | 142

5. Primary Outcome: Change in Self Reported Physical Recovery
Description: As determined using the Physical Component Score of Short form (SF) SF-36. Score range: 0-100, higher scores indicate a better health state. The change was determined between baseline and 6 months.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMH Intervention | Usual Care
Number analyzed (Participants) | 158 | 165
score on a scale | 36.86 (12.53) | 38.04 (12.09)

6. Primary Outcome: Change in Physical Recovery
Description: As determined using the Short Physical Performance Battery (SPPB). SPPB total score ranges from 0 (worst performance) to 12 points (best performance). The change was determined between baseline and 6 months.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMH Intervention | Usual Care
Number analyzed (Participants) | 84 | 92
score on a scale | 7.02 (4.39) | 7.66 (3.91)

7. Primary Outcome: Change in Self Reported Psychological Recovery
Description: As determined using the Mental Component Score of SF-36. Score range: 0-100, higher scores indicate a better health state. The change was determined between baseline and 6 months.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMH Intervention | Usual Care
Number analyzed (Participants) | 158 | 165
score on a scale | 53.72 (10.22) | 53.01 (10.64)

8. Secondary Outcome: Change in Depression Symptoms
Description: As determined using the (Patient Health Questionnaire) PHQ-9. The scale is from 1 - 27 with higher scores related to worse depression severity. The change was determined between baseline and 12 months.
Time Frame: 12 months
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | TMH Intervention | Usual Care
Number analyzed (Participants) | 148 | 150
score on a scale | 4.31 (4.79) | 4.44 (5.58)

9. Secondary Outcome: Change in Anxiety Symptoms
Description: As determined using the (Generalized Anxiety Disorder) GAD-7. Scores range from 0-21, with higher scores indicating worse symptoms. The change was determined between baseline and 12 months.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMH Intervention | Usual Care
Number analyzed (Participants) | 148 | 151
score on a scale | 3.39 (4.36) | 3.61 (4.80)

10. Secondary Outcome: Cost Effectiveness
Description: As determined using the cost-effectiveness ratio
Time Frame: 6 and 12 months
Population: Financial data were not collected so we have not done this analysis.
Arm/Group | TMH Intervention | Usual Care
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change in Depression Symptoms
Description: As determined using the (Patient Health Questionnaire) PHQ-9. The scale is from 1 - 27 with higher scores related to worse depression severity. The change was determined between baseline and 6 months.
Time Frame: 6 months
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | TMH Intervention | Usual Care
Number analyzed (Participants) | 158 | 165
score on a scale | 4.73 (5) | 4.31 (4.62)

12. Secondary Outcome: Change in Anxiety Symptoms
Description: As determined using the (Generalized Anxiety Disorder) GAD-7. Scores range from 0-21, with higher scores indicating worse symptoms. The change was determined between baseline and 6 months.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMH Intervention | Usual Care
Number analyzed (Participants) | 157 | 166
score on a scale | 3.64 (4.36) | 3.60 (4.31)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | TMH Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 6/216 | 11/213
Serious Adverse Events (participants affected / at risk) | 0/216 | 0/213
Other Adverse Events (participants affected / at risk) | 0/216 | 0/213

LIMITATIONS AND CAVEATS:
One outcome measure, the SPPB, was only validated in face-to-face assessments but it had to be adapted for telehealth evaluation during the pandemic. Care coordinator visits switched from a combination of in person and remote to fully remote after the pandemic started.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/20/NCT03108820/Prot_SAP_000.pdf